CLINICAL TRIAL: NCT06976580
Title: Effect of Skin Stretching on Pain Reduction During Local Anesthetic Injections: A Randomized Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2025-0207
Record Dates: First submitted 2025-04-21; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spinal Stenosis With Bilateral Lower Extremity Radiculopathy
Keywords: skin stretching; local anesthetic injection pain; lumbar spinal stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): conventional local anesthetic group
  Interventions: Procedure: conventional local anesthetic injection
- skin stretching group (Active Comparator): skin stretching group for anesthetic local injection
  Interventions: Procedure: skin stetching technique for local anesthetic injection

INTERVENTIONS:
Procedure: conventional local anesthetic injection — A conventional infiltration anesthesia will be conducted on the lumbar area of the patient, targeting the epidermis and subcutaneous tissue. A 25G syringe will be used, with the needle angle set between 30° and 45°. 1cc of 1% lidocaine will be injected. The target size of the wheal is 5-10 mm.
  Arms: control group
Procedure: skin stetching technique for local anesthetic injection — Skin stretching techinique will be applied to the local anesthetic injection site by stretching the skin around the needle entry point.
  Arms: skin stretching group

SUMMARY:
The purpose of this study is to investigate the potential analgesic effect of skin stretching during local anesthetic injection in patients with chronic lumbar pain and bilateral lower extremity radiculopathy undergoing selective transforaminal nerve block. This research is based on the hypothesis that mechanical skin stretching can reduce injection-related pain by facilitating the dispersion of the anesthetic agent and decreasing tissue resistance. By comparing the skin stretching technique with the conventional method of local anesthetic administration, this study aims to evaluate differences in pain perception, discomfort, and behavioral pain responses. The ultimate goal is to provide evidence for a simple, non-invasive, and effective intervention that can improve patient comfort and enhance the quality of clinical pain management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older with chronic low back pain lasting for more than 3 months, accompanied by bilateral lower extremity radiculopathy, who require Selective Transforaminal Epidural Block (STEB).
* Patients with a Numerical Rating Scale (NRS) score of 5/10 or higher, with pain that affects daily life activities.

Exclusion Criteria:

* Patients whose pain is influenced by mechanisms other than radiculopathy, such as peripheral neuropathy or myelopathy.
* Patients with a history of lumbar surgery within the last 6 months, or spinal injection treatment within the last 3 months.
* Patients with a history of allergy to local anesthetics, steroids, or contrast agents, or those at increased bleeding risk due to anticoagulant use (INR > 1.2).
* Patients with localized infections, sepsis, uncontrolled diabetes, or hypertension.
* Patients who are unable to consent or cooperate with the study procedures (e.g., cognitive impairment, severe mental illness).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | immediately after the local injection
  A comparison of pain score between control (conventional local anesthetic method) and skin stretching group using NRS.

SECONDARY OUTCOMES:
unpleasantness score | immediately after for unpleasantness score, behavior pain score, and 1 month after for soreness, respectively.
  A comparison of unplesantness score(NRS), and skin stretching group.
behavior pain score | immediately after for unpleasantness score, behavior pain score, and 1 month after for soreness, respectively.
  pain behavior using Pain Assessment in Advanced Dementia (PAINAD) scale, and skin stretching group.
soreness around the injection site | immediately after for unpleasantness score, behavior pain score, and 1 month after for soreness, respectively.
  soreness around the injection site between control (conventional local anesthetic method) and skin stretching group using NRS (numeral rating scale).

IPD SHARING:
Plan to Share IPD: No